CLINICAL TRIAL: NCT00989248
Title: Comparative Study of Cardiopulmonary Exercise Test on Land and Underwater in Patients With Congestive Heart Failure
Brief Title: Comparative Study of Cardiopulmonary Exercise Test Land Versus Water
Acronym: CHF
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Mauricio Koprowski Garcia, Instituto de Medicina Física e Reabilitação - HC - FMUSP
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CAPPESq 0532/08
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Congestive Heart Failure
Keywords: Ergospirometry; Cardiopulmonary Exercise Test; Exercises; Immersion
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- comparation VE/VO2 and VE/VCO2 (Experimental)
  Interventions: Other: Aerobic and anaerobic capacity use aquatic exercises

INTERVENTIONS:
Other: Aerobic and anaerobic capacity use aquatic exercises — Improve aerobic capacity use aquatic exercises in patients with Congestive Heart Failure
  Other Names: Aerobic and anaerobic capacities

SUMMARY:
At the neck level immersion, the water pressure causes significant displacement of blood from the lower limbs to the Intrathoracic circulation, triggering adaptive physiological responses due to the increase in central blood volume and consequent cardiovascular burdens. Immersion in warm water breaks the homeostasis, stimulates regulation mechanisms and responses of organs and systems beneficial to healthy and heart failure individuals. In literature there are a growing number of studies demonstrating the efficacy of exercises performed in the water.

DETAILED DESCRIPTION:
This study is about to compare the responses of one effort in two different environment. A group of 90 men, age between 55 to 75 years old recruited after a medical consultation, with the diagnostic of Congestive Heart Failure (CHF), under treatment at the Institute of Medicine and Rehabilitation and Institute Dante Pazzanesi, considered clinically stable (no cardiac symptoms or changes in medication for at least 30 days) and Funcional Class I, II, III according to NYHA.

Experimental Design: Patients will perform an test, first on land, and in a week time in a underwater treadmill. The data will be collected in four distinct moments: 1- anaerobic threshold (AT), 2- respiratory compensation point (RCP), 3- maximal effort (ME) and recovery (R). We will compare the following variables: test total time; perceived exertion scale (Borg); Heart rate (HR); Oxygen consumption (VO2); Carbon Dioxide production (VCO2); Oxygen pulse (VO2/FC); the ventilatory efficiency (VE/VO2) and (VE/VCO2); Respiratory quotient (VCO2/VO2); Systolic and Diastolic blood pressure; electrocardiographic changes, compatible with ischemia or arrhythmia.

ELIGIBILITY:
Inclusion Criteria: Patientes, 55 - 75 year, with Congestive Heart Failure (CHF)Functional class I - II and III according to the New York Heart Association (NYHA) and Injection Fracion 32% to 38%

Exclusion Criteria: Any peripheral artery disease, diabetes, pulmonary disease, hypertension (blood pressure >160/90) or significant cardiovascular morbidity.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
To appraisal the cardiopulmonar activities during the effort on land and in immersion | one year

SECONDARY OUTCOMES:
To develop an especific water protocol for reabilitations of patients with Congestive Heart Failure (CHF). The authors expect a beneficial adaptive response to the exercise in water comparing exercise on land. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio K Garcia, PhD, Study Chair — Shool of Medicine, University of São Paulo
Locations (1):
- Clinical Hospital, School of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Garcia MK, Rizzo L, Yazbek-Junior P, Yutiyama D, Silva FJD, Matheus D, Mastrocolla LE, Massad E. Cardiorespiratory performance of coronary artery disease patients on land versus underwater treadmill tests: a comparative study. Clinics (Sao Paulo). 2017 Nov;72(11):667-674. doi: 10.6061/clinics/2017(11)04. PMID 29236912